CLINICAL TRIAL: NCT06077630
Title: Non-attendance to Pediatric Outpatient Appointments: Prevalence, Associated Factors and Prediction Models
Brief Title: Non-attendance Prediction Models to Pediatric Outpatient Appointments
Status: Completed | Type: Observational
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Principal Investigator, Mariano Esteban Ibarra, Staff Pediatrician, Hospital General de Niños Pedro de Elizalde
Other Study IDs: 4084
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Non-Attendance, Patient; No-Show Patients
MeSH Terms: conditions — No-Show Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Attended appointments: An appointment scheduled by a patient that was attended
  Interventions: Other: No intervention
- Not-attended appointments: An appointment scheduled by a patient that was not-attended, regardless of the cause
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention, observational study

SUMMARY:
Non-attendance to pediatric outpatient appointments is a frequent and relevant public health problem.

Using different approaches it is possible to build non-attendance predictive models and these models can be used to guide strategies aimed at reducing no-shows. However, predictive models have limitations and it is unclear which is the best method to generate them. Regardless of the strategy used to build the predictive model, discrimination, measured as area under the curve, has a ceiling around 0.80. This implies that the models do not have a 100% discrimination capacity for no-show and therefore, in a proportion of cases they will be wrong. This classification error limits all models diagnostic performance and therefore, their application in real life situations. Despite all this, the limitations of predictive models are little explored.

Taking into account the negative effects of non-attendance, the possibility of generating predictive models and using them to guide strategies to reduce non-attendance, we propose to generate non-attendance predictive models for outpatient appointments using traditional logistic regression and machine learning techniques, evaluate their diagnostic performance and finally, identify and characterize the population misclassified by predictive models.

ELIGIBILITY:
Inclusion Criteria:

* pediatric outpatient appointments

Exclusion Criteria:

* appointments generated for system benchmarking or appointments with missing data

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All scheduled pediatric outpatient appointments between January 1 2017 and 31 december 2018 will be included. The sample will be randomized to allocate a generation cohort (two-thirds of the sample) and a validation cohort (one third of the sample).
Sampling Method: Probability Sample
Enrollment: 300000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Predictive Model non-attendance discrimination | 12 months
  Area Under the ROC Curve
Predictive Model non-attendance calibration | 12 months
  Calibration chart with predicted vs observed probability.
Predictive Model non-attendance diagnostic performance | 12 months

SECONDARY OUTCOMES:
Characterize the appointments misclassified by predictive models (FP) | 12 months
  False positive appointments prevalence
Characterize the appointments misclassified by predictive models (FN) | 12 months
  False negative appointments prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Ibarra, MD, Mag, Principal Investigator — Hospital General de Niños Pedro de Elizalde; Diego H Giunta, MD, MPH, PhD, Principal Investigator — Hospital Italiano de Buenos Aires; Arda Yilal, Engineer, Principal Investigator — Karolinska Institutet; Leticia Peroni, MD, Mag, Principal Investigator — Hospital Italiano de Buenos Aires; Lucia Perez, MD, Principal Investigator — Hospital Italiano de Buenos Aires

IPD SHARING:
Plan to Share IPD: No